CLINICAL TRIAL: NCT04462718
Title: Analysis of the Efficacy in the Lomg Term (Six Months Follow up) of the Combination of Radiofrecuency and Therapeutic Exercise Versus Therapeutic Exercise Alone in the Treatment of Patellofemoral Pain Syndrome.
Brief Title: Efficacy Analysis in Long Term of Radiofrecuency Combined vs. T.E. in the Treatment of Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Manuel Albornoz Cabello, Clinical Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RvsTE6MFU
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Musculoskeletal; Physical Medicine / Rehabilitation; Physiotherapy; Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with unilateral or bilateral PFPS will be divided into two groups, randomly selected (experimental group and control group), of 45 subjects each.
  Allocation was concealed and it was done by central randomisation by computer (EPIDARcomputer program).
  The subjects of the experimental group will undergo a program of supervised physical therapeutic exercise. And the subjects of the control group will follow the medical-pharmacological treatment and the ergonomic recommendations according to the established protocol.
  The target population will be all patients diagnosed with patellofemoral pain syndrome (PFPS) unilaterally or bilaterally, from the health area of La Rinconada while the eligible population will be composed of all those patients residing in or around Seville who can and wish to be part of it. of the study and that they meet the inclusion and exclusion criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP: (Active Comparator): You will be provided exclusively therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks.
  Interventions: Other: Therapeutic Exercise
- EXPERIMENTAL GROUP (Experimental): After the initial evaluation, the first 10 treatment sessions will be developed at the rate of five daily sessions in the first week, three sessions on alternate days in the second week and two sessions on alternate days in the third week (3 weeks in total), applying the monopolar capacitive diathermy with radiofrequency in the anterior aspect of the knee, in dynamic application in one of the members: affect or randomized (uni or bilateral pathology, respectively). This diathermy will be combined with a therapeutic exercise program supervised by a Physiotherapist.
  The treatment is administered with a pulsatile short-wave equipment and inductive electrodes of 100 W peak power, with a frequency of application of twice daily with a dose submitis (grade I), for 10 min, with a frequency of repetition of the impulses of 46 Hz and a pulse duration of 0.2 ms.
  Interventions: Other: Radiofrecuency

INTERVENTIONS:
Other: Radiofrecuency — EXPERIMENTAL GROUP: After the initial evaluation, the first 10 treatment sessions will be developed at the rate of five daily sessions in the first week, three sessions on alternate days in the second week and two sessions on alternate days in the third week (3 weeks in total), applying the monopolar capacitive diathermy with radiofrequency in the anterior aspect of the knee, in dynamic application in one of the members: affect or randomized (uni or bilateral pathology, respectively). This diathermy will be combined with a therapeutic exercise program supervised by a Physiotherapist.
  Arms: EXPERIMENTAL GROUP
Other: Therapeutic Exercise — CONTROL GROUP: will be provided exclusively therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks. They will be evaluated at the end of that period and six moths later in order to have at least three timepoints to evaluate.
  Arms: CONTROL GROUP:

SUMMARY:
The present study aims to promote research in the field of Physiotherapy, focusing on a health problem of maximum relevance, such as patellofemoral pain syndrome.

Although these treatments seem to be based on theoretical reasoning, the evidence for the efficacy of these interventions is not well established. Therefore, we select from among all the therapeutic tools available in physiotherapy, a procedure of therapeutic physical exercise.

Main objectives:

To know the efficacy of a therapeutic physical exercise protocol in the reduction of pain and the improvement of functional disability in patients with patellofemoral pain syndrome (PFPS).

Secondary objectives:

* Quantify the reduction of pain in the anterior aspect of the knee in patients with patellofemoral pain syndrome (PFPS), after treatment with monopolar capacitive diathermy by radiofrequency.
* To evaluate the improvement of functional disability in patients with patellofemoral pain syndrome (PFPS), after treatment with monopolar capacitive diathermy by radiofrequency.

Study hypothesis:

The treatment of patellofemoral pain syndrome (PFPS) with a therapeutic physical exercise protocol produces statistically significant changes in the reduction of pain and functional disability and the normalization of the anthropometric values of the joint balance of the knee

DETAILED DESCRIPTION:
At first, a meeting will be held with the patients under study where they will be informed and any doubts that may arise in relation to the investigation will be resolved. In addition, the correct adaptation of these to the inclusion and exclusion criteria of our study will be verified. Subsequently, they will be given individually the informed consent prepared expressly for the present study, the doubts arising with respect to this one will be resolved and their signature will proceed. At this time, and individually again, we will proceed to the development of the Clinical History of Physiotherapy where only the information necessary for our study will be collected.

To emphasize in this point that the participants will grant their consent for the treatment of the data obtained for scientific purposes, according to the legal norms.

Next, the patients will be randomly assigned to two groups: control group and experimental group. The randomization of the sample was done through the EPIDAR software in version 3.1 between the Experimental Group and the Control Group Subsequently, the evaluations and measurements of the study variables will be carried out by the research team.

CONTROL GROUP: You will be provided exclusively therapeutic exercises protocol to develop supervised by Physical Therapist that you must perform following a daily activity for three weeks. They will be evaluated at the end of that period and six moths later in order to have at least three timepoints to evaluate.

EXPERIMENTAL GROUP: After the initial evaluation, the first 10 treatment sessions will be developed at the rate of five daily sessions in the first week, three sessions on alternate days in the second week and two sessions on alternate days in the third week (3 weeks in total), applying the monopolar capacitive diathermy with radiofrequency in the anterior aspect of the knee, in dynamic application in one of the members: affect or randomized (uni or bilateral pathology, respectively). This diathermy will be combined with a therapeutic exercise program supervised by a Physiotherapist.

The treatment is administered with a Diathermy equipment and inductive electrodes of 100 W peak power, with a frequency of application of twice daily with a dose submitis (grade I), for 10 min, with a frequency of repetition of the impulses of 46 Hz and a pulse duration of 0.2 ms

After the tenth treatment session all the measurements will be repeated following the same environmental conditions as at the beginning and by the evaluators themselves to the components of both groups.Those measurements will be evaluated at the end of that three weeks period and six moths later in order to have at least three timepoints to evaluate.

ELIGIBILITY:
Inclusion Citeria:

1. Age from 18 to 55
2. . Patients with anterior knee pain were referred by a primary care physician at a public health center in southern Spain. Those participants with a self-reported pain intensity = 30 mm on the Visual Analog Scale (VAS) and a score <45 points in personal psychology The Apprehension Scale (PPAS) were invited to participate. The PPAS is a valid, reliable and easy-to-use tool for assessing the apprehension of subjects to receive electrical stimulation therapy.

Exclusion Criteria:

1. Any contraindication for the use of MDR.
2. Present cognitive alterations.
3. Have undergone conservative or surgical treatment of the knee in less than 6 months.
4. Having received injections of corticosteroids or hyaluronic acid; impaired cognition or communication; and be involved in an ongoing medical-legal dispute.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The perception of pain through the Visual Analogue Scale (EVA). | Time point 1: before the intervention
  The perception of pain through the Visual Analogue Scale (EVA). This variable has been obtained through a validated scale of 10 centimeters (0-10), where the subject self-positioned from absence of pain to the worst bearable pain.
The perception of pain through the Visual Analogue Scale (EVA). | Time point 2: when the intervention was finished (after 10 sesions : 2 weeks)
  The perception of pain through the Visual Analogue Scale (EVA). This variable has been obtained through a validated scale of 10 centimeters (0-10), where the subject self-positioned from absence of pain to the worst bearable pain.
The perception of pain through the Visual Analogue Scale (EVA). | Time point 3: six months later the initial evaluation.
  The perception of pain through the Visual Analogue Scale (EVA). This variable has been obtained through a validated scale of 10 centimeters (0-10), where the subject self-positioned from absence of pain to the worst bearable pain.
Kujala Score. | Time point 1: before the intervention
  The functional disability, quantified by means of the tests: Kujala Score.
Kujala Score. | Time point 2: when the intervention was finished (after 10 sesions : 2 weeks)
  The functional disability, quantified by means of the tests: Kujala Score.
Kujala Score. | Time point 3: six months later the initial evaluation.
  The functional disability, quantified by means of the tests: Kujala Score.

SECONDARY OUTCOMES:
Active and Pasive Knee's Range of Movement | Time point 1: before the intervention.
  In addition an anthropometric study of knee joint range of movement will be performed. Evaluating the Active and Pasive Knee's Range of Movement using universal goniometer measurement. we pay special attention to the possible restrictions in the normal range of motion
Active and Pasive Knee's Range of Movement | Time point 2: when the intervention was finished (after 10 sesions : 2 weeks)
  In addition an anthropometric study of knee joint range of movement will be performed. Evaluating the Active and Pasive Knee's Range of Movement using universal goniometer measurement. we pay special attention to the possible restrictions in the normal range of motion
Active and Pasive Knee's Range of Movement | Time point 3: six months later the initial evaluation.
  In addition an anthropometric study of knee joint range of movement will be performed. Evaluating the Active and Pasive Knee's Range of Movement using universal goniometer measurement. we pay special attention to the possible restrictions in the normal range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Cristo Jesús Barrios Quinta, Seville, Spain

IPD SHARING:
Plan to Share IPD: No